CLINICAL TRIAL: NCT01475097
Title: A Phase 4 Randomized, Double-blind Study Comparing Patient Comfort and Safety Between Iodixanol 320 mg I/mL and Iopamidol 370 mg I/mL in Patients Undergoing Peripheral Arteriography
Brief Title: Comparing Patient Comfort and Safety Between Iodixanol and Iopamidol in Patients Undergoing Peripheral Arteriography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: i3 Statprobe (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GE-012-098
Record Dates: First submitted 2011-11-03; First posted 2011-11-21 (Estimated); Results first posted 2014-04-15 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Drug Safety
Keywords: AE - Adverse event; Arteriography; IA - Intra-arterial; IOCM - Iso-Osmolar Contrast Medium; LOCM - Low-Osmolar Contrast Medium; Patient Comfort; Body Image Disturbance; Patient
MeSH Terms: interventions — iodixanol; Iopamidol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Arm (Active Comparator)
  Interventions: Drug: Iodixanol
- Comparator Arm (Active Comparator)
  Interventions: Drug: Iopamidol

INTERVENTIONS:
Drug: Iodixanol — Iodixanol 320 mg I/mL given by intra-arterial administration. Comparator agent Isovue (iopamidol) 370 mg I/mL given as intra-arterial administration.
  Other Names: Visipaque
  Arms: Active Arm
Drug: Iopamidol — Iodixanol 320 mg I/mL given by intra-arterial administration. Comparator agent Isovue (iopamidol) 370 mg I/mL given as intra-arterial administration.
  Other Names: Isovue
  Arms: Comparator Arm

SUMMARY:
The purpose of this study is to evaluate and compare overall patient comfort profile between an Iso-osmolar contrast media (IOCM), iodixanol 320 mg I/mL, and a Low-osmolar contrast media (LOCM), iopamidol 370 mg I/mL in patients undergoing arteriography of peripheral arteries.

ELIGIBILITY:
Inclusion Criteria:

* The subject is over 18 years old.
* Subjects are referred to undergo a peripheral arteriography as part of their routine clinical care.

Exclusion Criteria:

* The subject has known allergies to iodine or any prior history of adverse reaction to iodinated CM.
* The subject received another administration of CM within 24 hours prior to baseline or is scheduled to receive one within the 24 hour follow-up period.
* The subject is pregnant or lactating.
* The subject is taking metformin (e.g., Glucophage®) but is not willing or unable to discontinue at the time of the study procedure.
* The subject manifests thyrotoxicosis or is on dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Lim, PharmD, Study Director — GE Healthcare
Locations (1):
- GE Healthcare, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 255 subjects were enrolled in this study. Two (2) subjects did not complete the study. Total number of subjects that completed the study was 253.
Pre-assignment Details: Total of 255 subjects enrolled in this study. 2 subjects discontinued the study prior to contrast administration. Therefore, 253 subjects completed the study.
Groups:
- Iodixanol 320mgI/mL: Iodixanol 320 mg I/mL given by intra-arterial administration. Comparator agent Isovue (iopamidol) 370 mg I/mL given as intra-arterial administration.
- Iopamidol 370mgI/mL: Comparator agent Isovue (iopamidol) 370 mg I/mL given as intra-arterial administration.
Period: Overall Study
Arm/Group | Iodixanol 320mgI/mL | Iopamidol 370mgI/mL
Started | 128 | 127
Completed | 127 | 126
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iodixanol 320mgI/mL | Iopamidol 370mgI/mL | Total
Number analyzed (Participants) | 127 | 126 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (13.34) | 62.0 (15.30) | 63.2 (14.38)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 68 | 123
  >=65 years | 72 | 58 | 130
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 45 | 94
  Male | 78 | 81 | 159
Region of Enrollment [Number; unit: participants]
  United States | 27 | 24 | 51
  Germany | 38 | 39 | 77
  Spain | 57 | 58 | 115
  United Kingdom | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Subjects Experiencing Discomfort When Undergoing Peripheral Arteriography
Description: The number of subjects experiencing overall discomfort, heat or pain between Iodixanol and Iopamidol during the diagnostic phase of imaging.
Time Frame: Within 10 minutes post contrast administration.
Population: 249 subjects completed assessments, for overall discomfort, heat or pain between Iodixanol and Iopamidol during the diagnostic phase of imaging.124 subjects received Iodixanol and 125 subjects received Iopamidol.
Measure: Number; unit: participants
Arm/Group | Iodixanol 320mgI/mL | Iopamidol 370mgI/mL
Number analyzed (Participants) | 124 | 125
participants
  Discomfort | 53 | 92
  Heat | 48 | 82
  Pain | 5 | 21

2. Secondary Outcome: Comparison of Overall Image Quality Between Iodixanol and Iopamidol in Patients Undergoing Peripheral Arteriography.
Description: Overall Image Quality rated as 'Excellent, Adequate or Poor' by radiologists blinded to the contrast administration.
Time Frame: Within 10 minutes post contrast administration.
Population: A recruitment error occurred with a subject in each treatment group. Therefore, the subject's efficacy data were excluded from this efficacy analysis.
  This resulted in a total of 126 Iodixanol subjects and a total 125 Iopamidol subjects were used in the imaging analysis.
Measure: Number; unit: participants
Arm/Group | Iodixanol 320mgI/mL | Iopamidol 370mgI/mL
Number analyzed (Participants) | 126 | 125
participants
  Excellent | 109 | 103
  Adequate | 16 | 19
  Poor | 1 | 3

ADVERSE EVENTS:
Arm/Group | Iodixanol 320mgI/mL | Iopamidol 370mgI/mL
Serious Adverse Events (participants affected / at risk) | 2/127 | 2/126
Other Adverse Events (participants affected / at risk) | 15/127 | 3/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iodixanol 320mgI/mL (N=127) | Iopamidol 370mgI/mL (N=126)
Acute Myocardial Infarction (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Vessel Puncture Site Hematoma (General disorders) | 1 (1) | 0 (0)
Retroperitoneal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemorrhage from femoral common artery (Vascular disorders) | 0 (0) | 1 (1)
Hypovolemic Shock (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iodixanol 320mgI/mL (N=127) | Iopamidol 370mgI/mL (N=126)
Photopsia (Eye disorders) | 7 (7) | 1 (1)
Dizziness (Nervous system disorders) | 8 (8) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No